CLINICAL TRIAL: NCT01211405
Title: Randomized, Triple-Blind, Phase 2 Pilot Study Comparing 3 Different Doses of MDMA in Conjunction With Manualized Therapy in 24 Veterans, Firefighters and Police Officers With Chronic Posttraumatic Stress Disorder (PTSD)
Brief Title: Study Comparing Three Doses of MDMA Along With Therapy in Veterans With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-8
Record Dates: First submitted 2010-08-06; First posted 2010-09-29 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: MDMA; Therapy; Veterans; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Low dose MDMA-assisted therapy (Active Comparator): Participants will receive 30 mg midomafetamine HCl (MDMA) with therapy during each of two blinded experimental sessions.
  Interventions: Drug: Low dose MDMA-assisted therapy; Behavioral: Therapy
- Medium dose MDMA-assisted therapy (Active Comparator): Participants will receive 75 mg midomafetamine HCl (MDMA) with therapy on each of two blinded experimental sessions.
  Interventions: Drug: Medium dose MDMA-assisted therapy; Behavioral: Therapy
- Full dose MDMA-assisted therapy (Experimental): Participants will receive 125 mg midomafetamine HCl (MDMA) with therapy during each of two blinded experimental sessions, followed by a third open label session.
  Interventions: Drug: Full dose MDMA-assisted therapy; Behavioral: Therapy

INTERVENTIONS:
Drug: Low dose MDMA-assisted therapy — 30 mg midomafetamine HCl administered p.o. once at start of an experimental session. Upon mutual agreement, this may be followed by a supplemental dose of 15 mg 1.5 to 2 hours later
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine; midomafetamine
  Arms: Low dose MDMA-assisted therapy
Drug: Medium dose MDMA-assisted therapy — 75 mg midomafetamine HCl administered p.o. once at start of an experimental session. Upon mutual agreement, this may be followed by a supplemental dose of 37.5 mg 1.5 to 2 hours later
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine; midomafetamine
  Arms: Medium dose MDMA-assisted therapy
Drug: Full dose MDMA-assisted therapy — 125 mg midomafetamine HCl administered p.o. once at start of an experimental session. Upon mutual agreement, this may be followed by a supplemental dose of 62.5 mg 1.5 to 2 hours later
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine; midomafetamine
  Arms: Full dose MDMA-assisted therapy
Behavioral: Therapy — Non-directive therapy during each session

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective and reducing PTSD symptoms in veterans with chronic PTSD. The main question it aims to answer is: Do three doses of MDMA reduce PTSD symptoms?

Researchers will compare 30, 75, and 125 mg of MDMA HCl with therapy to see which dose best reduces PTSD symptoms.

Participants will undergo three preparatory non-drug therapy sessions with a male and female co-therapist team, then undergo three day-long MDMA-assisted therapy sessions after receiving an initial dose of 30, 75, or 125 mg MDMA HCl. After each MDMA-assisted therapy session, participants will undergo three integrative therapy sessions.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, dose comparison study with an open-label cross-over segment that will assess the safety and efficacy of MDMA-assisted therapy in veterans with chronic PTSD. Twelve of 24 participants will receive the full dose of 125 mg, six will receive 75 mg and six will receive 30 mg (active placebo dose) of MDMA HCl. An independent rater blind to condition will assess symptoms of PTSD and depression, general quality of life and posttraumatic growth prior to any therapy sessions one month after the second experimental session.

After undergoing three 90-minute non-drug introductory therapy sessions with a male/female co-therapist team, study participants will undergo two eight-hour long experimental sessions scheduled three to five weeks apart, prior to which they will be randomized to receive an initial dose of 30, 75 or 125 mg MDMA HCl , followed by a supplemental dose of half the initial dose 1.5 to 2.5 hours later. Participants will undergo integrative therapy in between each experimental session, including on the day after each session. Vital signs and psychological distress will be measured throughout each experimental session, and suicidality will be assessed throughout the course of the study. Spontaneously reported side effects will be collected on the day of each experimental session, and for six days afterward. PTSD symptoms, symptoms of depression, general psychological function, posttraumatic growth and quality of sleep will be assessed one month after the second experimental session, and the blind will be broken.

Participants who received 125 mg MDMA HCl will continue to have a third experimental session, and they will be assessed two months after the third experimental session.

Participants who received 30 or 75 mg MDMA HCl may take part in an open-label crossover segment that will follow nearly identical procedures, except that there will only be one introductory session prior to the first experimental session. There will be three experimental sessions. Symptoms of PTSD, depression and posttraumatic growth will be assessed at the start of the study. They will also be assessed one month after the second and two months after the third experimental session.

All participants will be assessed 12 months after their final experimental session. PTSD and depression symptoms and posttraumatic growth will be assessed, and participants will complete a questionnaire concerning the costs and benefits of being in the study.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with chronic PTSD, duration of 6 months or longer resulting from traumatic experience during military service;
* Have a CAPS score showing moderate to severe PTSD symptoms;
* Have had at least one unsuccessful attempt at treatment for PTSD either with talk therapy or with drugs, or discontinuing treatment because of inability to tolerate psychotherapy or drug therapy.
* Are at least 18 years old;
* Must be generally healthy;
* Must sign a medical release for the investigators to communicate directly with their therapist and doctors;
* Are willing to refrain from taking any psychiatric medications during the study period;
* Willing to follow restrictions and guidelines concerning consumption of food, beverages, and nicotine the night before and just prior to each experimental session;
* Willing to remain overnight at the study site;
* Agree to have transportation other than driving themselves home or to where they are staying after the integrative session on the day after the MDMA session;
* Are willing to be contacted via telephone for all necessary telephone contacts;
* Must have a negative pregnancy test if able to bear children, and agree to use an effective form of birth control;
* Must provide a contact in the event of a participant becoming suicidal;
* Are proficient in speaking and reading English;
* Agree to have all clinic visit sessions recorded to audio and video
* Agree not to participate in any other interventional clinical trials during the duration of this study.

Exclusion Criteria:

* Are pregnant or nursing, or if a woman who can have children, those who are not practicing an effective means of birth control;
* Weigh less than 48 kg;
* Are abusing illegal drugs;
* Have used ecstasy (material representing itself as MDMA) more than 5 times or at least once in the last 6 months;
* Are unable to give adequate informed consent;
* Upon review of past and current drugs/medication must not be on or have taken a medication that is exclusionary;
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2016-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mithoefer, MD, Principal Investigator — Private Practice
Locations (1):
- Offices of Michael Mithoefer, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified outcome data appearing in any published reports upon request. IPD may include de-identified baseline, demographic and outcome measure data. To ensure participant privacy, it will never include PHI. Please contact the central trial contact for details about data sharing and data available.
Supporting Information: Study Protocol, SAP
Time Frame: Data and study-related documents will be available following primary publication of outcomes.
Access Criteria: Interested persons should correspond with the central contact for the study.

REFERENCES:
- [Result] Mithoefer MC, Mithoefer AT, Feduccia AA, Jerome L, Wagner M, Wymer J, Holland J, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. 3,4-methylenedioxymethamphetamine (MDMA)-assisted psychotherapy for post-traumatic stress disorder in military veterans, firefighters, and police officers: a randomised, double-blind, dose-response, phase 2 clinical trial. Lancet Psychiatry. 2018 Jun;5(6):486-497. doi: 10.1016/S2215-0366(18)30135-4. Epub 2018 May 1. PMID 29728331
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose MDMA (30 mg): Participants will receive 30 mg MDMA during each of two blinded experimental sessions.
  Low dose MDMA: 30 mg MDMA administered p.o. once during each experimental session. Upon mutual agreement this maybe followed by a supplemental dose of 15 mg MDMA 1.5 to 2 hours later
  Psychotherapy: Non-directive psychotherapy during each session
- Medium Dose MDMA (75 mg): Participants will receive 75 mg MDMA on each of two blinded experimental sessions
  Medium dose MDMA: 75 mg MDMA adminis5tered p.o. once at start of an experimental session. Upon mutual agreement, may be followed 1.5 to 2 hours later by a supplemental dose of 37.5 mg
  Psychotherapy: Non-directive psychotherapy during each session
- Full Dose MDMA (125 mg): Participants will receive 125 mg MDMA during each of two blinded experimental sessions, followed by a third open label session.
  Full dose MDMA: 125 mg MDMA administered p.o. at start of an experimental session. By mutual agreement, may be followed 1.5 to 2 hours later by a supplemental dose of 62.5 mg MDMA.
  Psychotherapy: Non-directive psychotherapy during each session
Period: Overall Study
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Started | 7 | 7 | 12
Completed Primary Endpoint | 7 | 7 | 12
Completed Stage 1 | 6 | 6 | 12
Completed Stage 2 | 6 | 6 | 0
Completed (Completed 12-month follow-up) | 6 | 7 | 11
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg) | Total
Number analyzed (Participants) | 7 | 7 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.7) | 29.1 (4.0) | 40.7 (11.1) | 37.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 7
  Male | 5 | 6 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White/Caucasian | 6 | 4 | 12 | 22
  Ethnicity: Latino/Hispanic | 1 | 1 | 0 | 2
  Ethnicity: Native American | 0 | 1 | 0 | 1
  Ethnicity: Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS-IV) From Baseline to Primary Endpoint
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 7 | 7 | 12
score on a scale | -11.4 (12.7) | -58.3 (9.8) | -44.3 (28.7)

2. Secondary Outcome: Change in Global Assessment of Function (GAF) From Baseline to Primary Endpoint
Description: The Global Assessment of Functioning (GAF) Scale is a numeric scale ranging from 0 through 100 that is used by mental health clinicians and physicians to subjectively rate the social, occupational, and psychological functioning of adults. Higher scores indicate better functioning.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 7 | 7 | 12
score on a scale | 1.1 (4.6) | 19.4 (6.1) | 18.4 (14.4)

3. Secondary Outcome: Change in Posttraumatic Growth Inventory (PTGI) From Baseline to Primary Endpoint
Description: The Posttraumatic Growth Inventory (PTGI) is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains five subscales; relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life. Questions are answered on a scale from 0 (I did not experience this change) to 5 (I experienced this change to a great degree). Items are added to calculate the total PTGI score which ranges from 0 to 105, with higher scores indicative of greater growth.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 7 | 7 | 12
score on a scale | -11.6 (12.2) | 36.1 (12.0) | 33.7 (24.0)

4. Secondary Outcome: Change in Beck Depression Inventory (BDI-II) From Baseline to Primary Endpoint
Description: Validated self-report measure of symptoms of depression. The BDI-II total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depressive symptoms. The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 7 | 7 | 12
score on a scale | -4.6 (8.8) | -15.4 (9.5) | -24.6 (10.6)

5. Secondary Outcome: Change in Dissociative Experience Scale (DES-II) From Baseline to Primary Endpoint
Description: The DES-II is a 28-item self-report measure of dissociation, defined as a lack of normal integration of an individual's thoughts, feelings, or experiences into the stream of consciousness or memory. Respondents indicate how often the specific experience happens to them, from "never" (0% of the time) to "always" (100%). The scale is scored by treating percentages as single digits and summing to produce a total score, ranging from 0 to 100. The higher the score, the more dissociative symptoms.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat [Note: The DES-II was added as an outcome measure in Protocol Amendment 5 so was not collected in participants who completed the study under an earlier version of the protocol (n=14).]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 3 | 3 | 6
score on a scale | 1.8 (0.95) | -8.6 (1.9) | -8.8 (6.2)

6. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline to Primary Endpoint
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. It is comprised of 18 items that yield seven component scores. Component scores are summed to create a total score. Total scores range from 0 (better) to 21 (worse), with higher scores indicating poor sleep quality.
Time Frame: Baseline to one month after second experimental session
Population: Intent-to-treat [Note: The PSQI was added as an outcome measure in Protocol Amendment 3 so was not collected in participants who completed the study under an earlier version of the protocol (n=6).]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose MDMA (30 mg) | Medium Dose MDMA (75 mg) | Full Dose MDMA (125 mg)
Number analyzed (Participants) | 5 | 5 | 10
score on a scale | 1.8 (2.8) | -6.4 (7.1) | -4.8 (4.1)

ADVERSE EVENTS:
Time Frame: During entire study duration (approx 12 months)
Groups:
- Blinded Low Dose MDMA-assisted Therapy: Participants will receive 30 mg midomafetamine HCl with therapy during each of two blinded experimental sessions.
- Blinded Medium Dose MDMA-assisted Therapy: Participants will receive 75 mg midomafetamine HCl with therapy on each of two blinded experimental sessions
- Blinded Full Dose MDMA-assisted Therapy: Participants will receive 125 mg midomafetamine HCl with therapy during each of two blinded experimental sessions, followed by a third open label session.
- Open-Label Low Dose MDMA-assisted Therapy: Participants who received two sessions of blinded low dose MDMA-assisted therapy were given the option to cross over and receive three additional open-label MDMA-assisted therapy sessions with 100 mg of midomafetamine HCl
- Open-Label Medium Dose MDMA-assisted Therapy: Participants who received two sessions of blinded medium dose MDMA-assisted therapy were given the option to cross over and receive three additional open-label MDMA-assisted therapy sessions with 100 mg of midomafetamine HCl
- Open-Label Full Dose MDMA-assisted Therapy: Participants who received two sessions of blinded full dose MDMA-assisted therapy received a third open-label session with 125 mg midomafetamine HCl
- Low Dose Group 12 Month Follow-Up; Medium Dose Group 12 Month Follow-Up; Full Dose Group 12 Month Follow-Up: Participants followed for 12 months from end of Stage or 2
- SRRS: Low Dose; SRRs: Medium Dose; SRRs: Full Dose: Spontaneously reported reactions (SRRs) on day of blinded experimental sessions and 7 days after.
Arm/Group | Blinded Low Dose MDMA-assisted Therapy | Blinded Medium Dose MDMA-assisted Therapy | Blinded Full Dose MDMA-assisted Therapy | Open-Label Low Dose MDMA-assisted Therapy | Open-Label Medium Dose MDMA-assisted Therapy | Open-Label Full Dose MDMA-assisted Therapy | Low Dose Group 12 Month Follow-Up | Medium Dose Group 12 Month Follow-Up | Full Dose Group 12 Month Follow-Up | SRRS: Low Dose | SRRs: Medium Dose | SRRs: Full Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/12 | 0/6 | 0/6 | 0/12 | 0/6 | 0/7 | 0/11 | 0/7 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 0/12 | 1/6 | 0/6 | 0/12 | 1/6 | 1/7 | 0/11 | 0/7 | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 6/7 | 4/7 | 8/12 | 6/6 | 4/6 | 4/12 | 0/6 | 0/7 | 0/11 | 7/7 | 7/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Low Dose MDMA-assisted Therapy (N=7) | Blinded Medium Dose MDMA-assisted Therapy (N=7) | Blinded Full Dose MDMA-assisted Therapy (N=12) | Open-Label Low Dose MDMA-assisted Therapy (N=6) | Open-Label Medium Dose MDMA-assisted Therapy (N=6) | Open-Label Full Dose MDMA-assisted Therapy (N=12) | Low Dose Group 12 Month Follow-Up (N=6) | Medium Dose Group 12 Month Follow-Up (N=7) | Full Dose Group 12 Month Follow-Up (N=11) | SRRS: Low Dose (N=7) | SRRs: Medium Dose (N=7) | SRRs: Full Dose (N=12)
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Low Dose MDMA-assisted Therapy (N=7) | Blinded Medium Dose MDMA-assisted Therapy (N=7) | Blinded Full Dose MDMA-assisted Therapy (N=12) | Open-Label Low Dose MDMA-assisted Therapy (N=6) | Open-Label Medium Dose MDMA-assisted Therapy (N=6) | Open-Label Full Dose MDMA-assisted Therapy (N=12) | Low Dose Group 12 Month Follow-Up (N=6) | Medium Dose Group 12 Month Follow-Up (N=7) | Full Dose Group 12 Month Follow-Up (N=11) | SRRS: Low Dose (N=7) | SRRs: Medium Dose (N=7) | SRRs: Full Dose (N=12)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hordeolum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venomous sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tic (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trichotillomania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 10
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abcess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep deficit (Nervous system disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 10
Depressed mood (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flashback (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 3 | 10
Intrusive thoughts (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Time perception altered (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudofolliculitis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypnopompic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Difficulty Concentrating (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
Dizziness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Drowsiness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Mouth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 7
Impaired Judgment (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Impaired Gait/Balance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 6
Jaw Clenching, Tight Jaw (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Lack of Appetite (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 6
Low Mood (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Muscle Tension (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 7
Need More Sleep (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 9
Perspiration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ruminations (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Sensitivity to Cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Weakness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2013-08-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT01211405/Prot_003.pdf
  • Statistical Analysis Plan (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT01211405/SAP_001.pdf
  • Informed Consent Form (2013-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT01211405/ICF_002.pdf